CLINICAL TRIAL: NCT01054040
Title: The Impact of Portion Plates for Weight Loss on Cardiac Rehabilitation Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Richmond Health Services (Other Government)
Responsible Party: Mary Flesher, Richmond Health Services
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H09-03467 (UBC Ethics Board)
Record Dates: First submitted 2010-01-20; First posted 2010-01-22 (Estimated); Last update posted 2010-01-22 (Estimated); Status verified 2010-01

CONDITIONS: Cardiovascular Disease
Keywords: cardiovascular disease, portion plate
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Standard nutrition cardiac care (No Intervention): Patients will receive standard care of group nutrition counselling and individual counselling if requested
  Interventions: Other: Portion plate given to cardiac rehabilitation patients

INTERVENTIONS:
Other: Portion plate given to cardiac rehabilitation patients — Patients in the experimental group will be provided with standard care (group and individual nutrition counselling) plus be provided a portion control plate
  Other Names: Divided portion control plate from StepsCount

SUMMARY:
The study will involve cardiac rehabilitation clients and will measure their weight, height, waist circumference and blood pressure comparisons between first and final visit (after 8 weeks). A control group will receive usual care and an experimental group will receive usual care plus a portion control plate for their meals. Patients currently have their waist circumference, weight, height and blood pressure measured at their first visit (week 0) and at their final visit (week 8). This study would compare these three parameters at these same times (week 0 and week 8) between the control and experimental groups. The control group would receive the usual care while the experimental group would receive usual care plus be given a portion control plate at week 0.

The hypothesis of this study is that subjects from the experimental group will have an average reduction in: (a) waist circumference by > 5%, (b) weight or BMI by > 5%, and (c) systolic and diastolic blood pressure by >10%. The subjects in the control group are hypothesized to show an average less than these targets for the experimental group.

DETAILED DESCRIPTION:
In Canada, 6.8 million adults are overweight and an additional 4.5 million are obese, which translates to about 58.3% of Canadian adults being overweight or obese. The overall cost of obesity in British Columbia (2006) is estimated to be $563 million dollars. An increase in food portion sizes and sedentary lifestyle of Canadians has contributed to the imbalance in caloric intake and usage. Obesity is the leading risk factor for many chronic diseases and has been linked directly to an increased incidence of heart disease and hypertension.

Cardiac Rehabilitation (CR) Phase I involves the rehabilitation of patients with cardiac disease in an outpatient setting at the Richmond Hospital. It is an 8-week interdisciplinary program involving exercise, group education, and individual counselling. Currently, patients are referred by a cardiologist to the CR program and have parameters like their blood pressure and waist circumference measured at the first and final visits. Over the past year, the average change in blood pressure from the first to last day (after 8 weeks) was a reduction of 12.2 systolic blood pressure and 3.1 diastolic blood pressure. The average waist circumference changed by 0.88 cm. Patients are offered an optional individual visit with the dietitian and are required to attend a weekly nutrition education class.

Weight Loss with Portion Plates Portion sizes are essential in determining the amount of calories consumed at meal times. When larger portions are consumed, there is a greater amount of calories ingested. The Canadian Community Health Survey (2004) found that the average adult consumed about 2732 kilocalories daily, which is increased from the average of 2356 kilocalories in 1991.

One randomized controlled study looked at the impact of a portion control tool (portion plate) on the weight changes in diabetic patients and found a significantly greater weight loss in patients using the tool versus the control group. No other studies were found that measured the efficacy of these tools in cardiac patients.

Hypertension and Weight Reduction Body mass index (BMI) is a common tool used to compare height and weight, that is calculated by weight (kg) divided by height squared (m²). A person with an acceptable body weight has a BMI of 18.5-24.9 kg/ m². Obesity is defined as a BMI of 30 kg/ m². Increased body weight or a high BMI is a risk factor for hypertension. A reduction in BMI through non-pharmacological methods like caloric reduction and physical activity has significantly improved cardiac risk factors in some studies.

Routine physical activity has been shown to reduce blood pressure. Studies on blood pressure and exercise have showed improvements of 10-20%. Systolic blood pressure was reduced by 1.6 mm Hg systolic and 1.1 mm Hg diastolic for every 1 kg of weight lost in overweight patients. Studies demonstrated that a reduction of each 100 mmol/day of dietary sodium was associated with a decline of 5-7 mmHg/2.7 mmHg in hypertensive subjects. Based on the literature, the experimental group was hypothesized to have a reduction of 10% of both systolic and diastolic blood pressure (or a systolic decrease of 13 mm Hg or more, and diastolic reduction of 8 mm Hg or more) versus a <10% reduction in the control group.

Waist Circumference and Weight Loss Waist circumference that is indicative of an increased risk of diseases, including coronary heart disease is 88 cm for women and 102 cm for men. Reducing waist circumference through weight loss can lower a person's risks of hypertension and coronary heart disease. Using waist circumference in combination with BMI is useful in determining a person's health risks, especially if the person has a normal BMI but a high waist circumference. Elevations in both BMI and waist circumference are independent risk factors in heart disease, increasing the heart disease risk factors by 2-4 fold.

Purpose of the Study:

The purpose of this study is to determine if the use of a portion control tool (portion plate) could improve the waist circumference, weight loss and blood pressure of the patients within a cardiac rehabilitation program. If the tool is shown to statistically improve these outcomes when compared with a control group receiving usual care, the tool may be added to the usual care of these patients in the long term.

Objectives and Research Question This randomized controlled study will ask: How will portion control plates impact the weight, blood pressure and waist circumference of patients in a cardiac rehabilitation program?

ELIGIBILITY:
Inclusion Criteria:

* patients attending the cardiac rehab program who have a waist circumference of more than 102 cm (males) and 89 cm (females)

Exclusion Criteria:

* any patients with a waist circumference below the above levels

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2010-02; Primary Completion 2011-02 (Estimated); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
Reduce waist circumference by 5% or more in intervention group | 8 weeks

SECONDARY OUTCOMES:
Reduce weight or BMI by 5% or more in intervention group | 8 weeks
Reduce diastolic and systolic blood pressure by 10% or more in intervention group | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Monica Redekopp, BSN, PhD, Study Director — Richmond Health Services
Locations (1):
- Richmond Health Services, Cardiac Rehabilitation, Richmond, British Columbia, Canada